CLINICAL TRIAL: NCT07021794
Title: Effectiveness of Treating Post-COVID-19 Conditions (Long COVID) With the SARS-CoV-2 Specific Monoclonal Antibody, Sipavibart
Brief Title: SARS-CoV-2 Specific Monoclonal Antibody for Post-COVID-19 Conditions (Long COVID)
Acronym: Monoclonal
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nancy Klimas (Other)
Collaborators: Florida Department of Health (Other Government)
Responsible Party: Sponsor-Investigator, Nancy Klimas, Director, Institute for Neuro Immune Medicine, Nova Southeastern University
Organization: Nova Southeastern University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LongCovid Monoclonal Antibody
Record Dates: First submitted 2024-10-31; First posted 2025-06-15 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-06

CONDITIONS: Post-COVID / Long-COVID
Keywords: LongCOVID; Monoclonal antibody (mAb) therapy; Post-viral conditions
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Mycobacterium Infections, Nontuberculous

STUDY DESIGN:
Intervention Model Description: This placebo-controlled, randomized, blinded, two-arm phase II study will test the safety and potential efficacy of the targeted mAb, Sipavibart (formerly AZD3152) in 100 patients with Long COVID.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sipavibart (Experimental): Participants receive a single intramuscular dose of Sipavibart, 300 mg intramuscular and are then followed for a duration of six months.
  Interventions: Drug: Placebo
- Placebo (Placebo Comparator): Participants receive single dose of placebo (saline) indistinguishable from the active drug in appearance, and are then followed for a duration of six months.
  Interventions: Biological: Sipavibart

INTERVENTIONS:
Drug: Placebo — A single dose of placebo (saline) indistinguishable from the active drug in appearance
  Arms: Sipavibart
Biological: Sipavibart — A single intramuscular dose of Sipavibart, 300 mg
  Arms: Placebo

SUMMARY:
This placebo-controlled, randomized, blinded, two-arm phase II study will test the safety and potential efficacy of the targeted mAb, Sipavibart (formerly AZD3152) in patients with Long COVID.

DETAILED DESCRIPTION:
Acute COVID-19 infection can present differently among infected patients, with the infection ranging in symptom presentation from asymptomatic and mild symptomatology to severe illness. Common symptoms tied to a COVID-19 infection include fever, chills, cough, respiratory ailments (shortness of breath or difficulty breathing), fatigue, muscle and/or joint pain, headache, loss of taste or smell, sore throat, congestion, and/or gastrointestinal (GI) disturbances (nausea, vomiting, and/or diarrhea). In some patients, these symptoms are short-lived and span the length of the acute infection, while in many patients the symptoms can linger for an extended period. Early indications point to inflammation playing a key role in acute COVID-19 illness and severity, and may play a role in prolonged Long COVID(LC) symptom intolerance and long-term sequelae. Researchers have demonstrated the involvement of persistent inflammation, poor antiviral responses, and evidence of chronic viral reactivation.

More recently, studies have demonstrated that mAb targeting the spike (S) protein of the SARS-CoV-2 may not only be effective in treating acute COVID-19 infection, especially variants prior to Omicron (alpha, beta, and delta), but also may play a role in addressing Long COVID. This implies that mAb infusions likely target SARS-CoV-2, decreasing activity, and potentially addressing disease pathogenesis tied to its activation, shutting down negative implications of inflammation tied to viral activation. This study will employ a two-arm randomized design to evaluate the efficacy of the drug Sipavibart in individuals experiencing LC symptoms. Participants will undergo six months of follow up after receiving either one dose of Sipavibart or one dose of placebo. After completion of the 6-month follow up, an open-label extension phase will be added at month 6 (week 24), where subjects who continue to experience symptoms of long COVID (regardless of the blinded treatment assignment) could be eligible to receive one dose of Sipavibart in an open-label fashion.

ELIGIBILITY:
Inclusion Criteria:

An individual is eligible for inclusion if all of the following apply:

1. 18 to 70 years old,
2. Inciting event: Acute COVID documented by testing (PCR or antigen testing in a clinical setting).
3. Onset of COVID symptoms occurring on or prior to August 31st, 2023; and persistence of symptomatic expression of Long COVID (defined #6 below) for more than 3 months after COVID diagnosis.
4. Current symptomatic expression meets the case definition of ME/CFS.
5. PROMIS 29 score at screening of moderate to severe (≥60).
6. Meets National Academy of Sciences (NAS) criteria for Long COVID with the following provisions:

   1. Allowance for normal illnesses of aging, such as hypertension and diabetes, if the conditions are treated and are in demonstrable stable and acceptable ranges at the time of screening and assessment. Specifically, blood pressures < 150 systolic and 90 diastolic mmHg are required.
   2. Allowance of stable comorbid conditions common in post viral illness, such as fibromyalgia, irritable bowel, interstitial cystitis, dysautonomia that have not required hospitalization in the two years prior to recruitment.
7. Able to provide written consent to study. Agrees to participate in follow-up visits.

Subject Exclusion Criteria

An individual is ineligible to participate if any of the following apply:

1. Known active acute SARS-CoV-2 infection ≤ 4 weeks from consent.
2. Known severe anemia, defined as < 8 g/dL.
3. Known stroke that resulted in cognitive impairment within 3 months of enrollment.
4. Self-report of current treated or untreated major depression with psychotic or melancholic features, schizophrenia, bipolar disorder, delusional disorders, dementias of any type, or a history of CNS disorders that may affect cognitive function (i.e., epilepsy, stroke, brain tumor, multiple sclerosis, Parkinson's Disease, Alzheimer's disease), or substance abuse during the last two years, excluding cannabis products.
5. Allergy to any ingredient of the study drug (self-report)

   1. Sipavibart is supplied as 150 mg/mL of active ingredient in 20 mM L-histidine/L-histidine hydrochloride, 220 mM L-arginine hydrochloride, and 0.04% (w/v) polysorbate 80, at pH 6.0.
   2. Hypersensitivity to other humanized mAbs.
6. Current heavy alcohol or tobacco use (self-report). Alcohol consumption not to exceed approximately 15 drinks per week (with a drink defined as 12 oz beer, 5 oz wine, or 1.5 oz distilled spirits) and tobacco use not to exceed 20 cigarettes (or equivalent) per day during the last month.
7. Active chronic infections such as HIV, Hepatitis B Virus (HBV), and Hepatitis C Virus (HCV), indicated by self-report, and abnormal liver function tests (>3x upper limit of normal) or evidence in the health record of chronic active hepatitis or human immunodeficiency virus (HIV).
8. Renal disease (self-report; laboratory results: renal insufficiency with serum creatinine > 2.0 mg/dL or eGFR < 44; or currently on renal dialysis)
9. Liver disease (self-report or laboratory results: hepatic insufficiency (bilirubin >2.5mg/dL or transaminases > 3X the upper limits of normal)
10. Uncontrolled diabetes, evidenced by combination of morning blood glucose and previous diagnosis of diabetes, AIC>7
11. Diagnosed with congestive heart failure or significant arrythmia (ventricular tachycardia with a rapid rate at rest (> 100 bpm), persistent atrial fibrillation, or second- or third-degree heart block)
12. Pre-existing sustained severe hypertension (BP >180/110 mmHg in the sitting position)
13. Any of the following within 4 weeks of consent (Self-reported/medical record):

    1. an acute myocardial infarction or unstable angina
    2. uncontrolled arrhythmias causing symptoms or hemodynamic compromise
    3. acute myocarditis or pericarditis, uncontrolled acutely decompensated heart failure (acute pulmonary edema)
    4. acute pulmonary embolism
    5. suspected dissecting aneurysm
    6. severe hypoxemia at rest
    7. any acute or chronic disorder that may affect exercise performance, or
    8. if they are aggravated by exercise (e.g., infection, thyrotoxicosis, unable to cooperate)
14. Diagnosed bleeding disorders or use of blood-thinning medications.
15. Current or previous receipt of any COVID antiviral medication within 30 days prior to screening (self reported)
16. Currently have exclusionary diagnoses that could reasonably explain the symptoms of their fatiguing illness and their severity, using the exclusion criteria best described in the Ambiguities in case definition paper for CFS, as described in detail in [13] which clarifies exclusionary conditions. These exclusionary diagnoses that are not otherwise listed above comprise:

    1. Organ failure
    2. Chronic inflammatory diseases
    3. Major neurologic diseases that could cause fatigue or neurologic deficits
    4. Diseases requiring systemic treatment (i.e., transplantation, chemotherapy, radiation)
    5. Major endocrine diseases
    6. Untreated primary sleep disorders
    7. BMI > 40 kg/m2
    8. Temporary conditions discovered at screening, such as

       * Temporary effects of medications
       * Temporary sleep deprivation
       * Untreated hypothyroidism, hypothyroidism that has been inadequately controlled during the last 3 months, or free T4 level not within normal limits
       * Active infection (for COVID-19 infection and other infections, participants may be rescreened six weeks after resolution of infection)
17. Known diagnosis of chronic Lyme disease with persistent symptoms, sequelae, or related therapy.
18. Any marijuana illicit drug use within 30 days of informed consent
19. Inability to discontinue symptomatic medications for the identified time periods
20. Moderate or severe immunocompromised patients, such as those described in the NIH COVID-Treatment Guidelines
21. Are scheduled for a surgery during the period of study participation, had minor surgery within three months prior to screening, or had major surgery within 6 months prior to screening
22. Participating in any interventional (including social-behavioral therapy) clinical trial of an investigational therapy within 6 weeks prior to consent, or planning to participate in another interventional clinical trial of an investigational therapy during the course of this study
23. COVID Vaccination within 90 days prior to entry and for the duration of the study
24. Pregnancy is excluded. Women of childbearing age will be given a pregnancy test.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System-29 | 12 weeks
  Comprehensive Symptom Burden Index (CSBI) total scores will serve as a composite outcome measure derived from eight PROMIS domains to capture overall symptom burden. Scores will be calculated at baseline and Week 12. Efficacy will be determined by the proportion of participants classified as IMPROVED, defined as having a ≥4.5-point increase in CSBI from baseline, a threshold representing moderate and clinically meaningful improvement.
Review of Treatment Related Adverse Events | 24 weeks
  Number of participants with treatment-related adverse events as assessed by frequency of safety events during the study period.

SECONDARY OUTCOMES:
Symptom-specific participant-reported outcome measures | 24 weeks
  Evaluate change in Comprehensive Symptom Burden Index (CSBI) score from baseline to Week 24 between Sipavibart and placebo groups.
Change in Simple Reaction Time (Milliseconds) | Baseline, 12 and 24 weeks
  Change in raw Simple Reaction Time, measured in milliseconds using the CNS Vital Signs computerized test battery, from baseline to Weeks 12 and 24.
Self-reported fatigue using MFI | 12 and 24 weeks
  Change in Multidimensional Fatigue Inventory (MFI) total and subscale scores (General Fatigue, Physical Fatigue, Mental Fatigue, Reduced Activity, Reduced Motivation) from baseline to Weeks 12 and 24.
  Correlation of MFI scores with PROMIS Fatigue and DSQ-PEM subscales (convergent validity).
Change in Heart Rate Post-6MWT | 12 and 24 weeks
  Change in Heart Rate post 6-minute walk distance (6MWT), in meters, from baseline to Weeks 12 and 24.Unit: Beats per minute (bpm)
Processing Speed | 12 and 24 weeks
  Change in Processing Speed score (Standard score or percentile) from baseline to Weeks 12 and 24 as measured by CNS Vital Signs.
Attention | Baseline, 12 and 24 weeks
  Change in Attention (Standard Score) from baseline to Weeks 12 and 24 as measured by CNS Vital Signs.
Systolic Blood Pressure Response During NASA Lean Test | Baseline, 12 and 24 Weeks
  Change in systolic blood pressure (mmHg) from baseline to 10 minutes upright during the NASA Lean Test
Diastolic Blood Pressure Response During NASA Lean Test | Baseline, 12 and 24 Weeks
  Change in diastolic blood pressure (mmHg) from baseline to 10 minutes upright during the NASA Lean Test
Symptom Score During NASA Lean Test | Baseline, 12 and 24 weeks
  Change in self-reported orthostatic intolerance symptom score, measured using a 0-10 numeric scale, during the NASA 10-minute Lean Test
Within-participant change in PROMIS Fatigue scores from baseline to Week 24 | Baseline, 12 weeks, 24 weeks
  PROMIS Fatigue domain score measured at baseline, Week 12, and Week 24 to assess change over time.
Within-participant change in PROMIS Pain Interference scores | Baseline, 12 weeks, 24 weeks
  PROMIS Pain Interference domain score measured at baseline, Week 12, and Week 24 to assess change over time.
Within-participant change in PROMIS Physical Function scores | Baseline, 12 weeks, 24 weeks
  PROMIS Physical Function domain score measured at baseline, Week 12, and Week 24 to assess change over time.
Change in PROMIS Cognitive Function 8a T-score | Baseline, 12 Week, 24 week
  Evaluates cognitive function using PROMIS Cognitive Function 8a at baseline, Week 12, and Week 24. Used to assess differential treatment effects by baseline symptom cluster (Cognitive Dysfunction group).
Change in Orthostatic Hypotension Questionnaire (OHQ) composite score | Baseline, 12 weeks, 24 weeks
  Evaluates autonomic dysfunction using the OHQ at baseline, Week 12, and Week 24. Used to assess differential treatment effects by baseline symptom cluster (Autonomic Dysfunction group).
Change in DePaul Symptom Questionnaire-Post-Exertional Malaise (DSQ-PEM) | Baseline, 12 weeks, 24 weeks
  Evaluates post-exertional malaise and exercise intolerance using the DSQ-PEM T score at baseline, Week 12, and Week 24. Used to assess differential treatment effects by baseline symptom cluster .
Change in DePaul Symptom Questionnaire (DSQ) score | Baseline, 12 weeks, 24 weeks
  Assesses symptom burden using the DSQ at baseline, Week 12, and Week 24.
Change in Pittsburgh Sleep Quality Index (PSQI) global score | Baseline, 12 weeks, 24 weeks
  Assesses sleep quality using the PSQI at baseline, Week 12, and Week 24. Scores (0-21)
Change in Brief Pain Inventory (BPI) severity score | Baseline, 12 weeks, 24 weeks
  Assesses pain severity using the BPI at baseline, Week 12, and Week 24. Scores (1-10).
Change in Modified Medical Research Council (mMRC) Dyspnea Scale score | Baseline, 12 weeks, 24 weeks
  Assesses dyspnea using the mMRC scale at baseline, Week 12, and Week 24. Score range 0-4
Change in Generalized Anxiety Disorder-7 (GAD-7) score | Baseline, 12 weeks, 24 weeks
  Assesses anxiety symptoms using the GAD-7 at baseline, Week 12, and Week 24. Score range 0-21
Change in Patient Health Questionnaire-8 (PHQ-8) score | Baseline, 12 weeks, 24 weeks
  Assesses depressive symptoms using the PHQ-8 at baseline, Week 12, and Week 24. Score range 0-24
Change in Brief Illness Perception Questionnaire (B-IPQ) total score | Baseline, 12 weeks, 24 weeks
  Assesses illness perception using the B-IPQ at baseline, Week 12, and Week 24. Score range 0-80
Change in Functional Capacity Scale (FUNCAP) score | Baseline, 12 weeks, 24 weeks.
  Assesses functional impairment using the FUNCAP scale at baseline, Week 12, and Week 24. Score range 0-100
Change in Composite Symptom Burden Index (CSBI) score | Baseline, 12 weeks, 24 weeks
  The CSBI is a derived score summarizing symptom burden across multiple validated domains (e.g., fatigue, pain, sleep, mood, cognitive function). Domain scores are standardized and averaged to produce a single CSBI value per participant. Paired differences from baseline to Week 12 and Week 24 will be analyzed to assess intra-individual changes and overall cohort-level trends.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Klimas, MD, Principal Investigator — Nova Southeastern University; Amanpreet Cheema, PhD, Study Director — Nova Southeastern University
Locations (1):
- Nova Southeastern University, Fort Lauderdale, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.nova.edu/nim/research-studies/long-covid.html